CLINICAL TRIAL: NCT00604708
Title: Observer Blinded, Randomized Phase 3 Study to Investigate the Non-Inferiority of IC51 vs. JE-VAX as Vaccines for Japanese Encephalitis in Healthy Subjects
Brief Title: Immunogenicity Study of the Japanese Encephalitis Vaccine IC51
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IC51-301
Record Dates: First submitted 2008-01-04; First posted 2008-01-30 (Estimated); Results first posted 2012-11-29 (Estimated); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IC51 (Experimental): 6 mcg (microgram) i.m. (intramuscular) on Day0, 14 and 28
  Interventions: Biological: IC51
- JE-VAX (Active Comparator): given s.c. on Day 0, 7 and 28
  Interventions: Biological: JE-VAX

INTERVENTIONS:
Biological: IC51 — IC51 (JE-PIV), 6 mcg, i.m. injection, 2 vaccinations, days 0 and 28
  Other Names: Japanese Encephalitis purified inactivated vaccine
  Arms: IC51
Biological: JE-VAX — JE-VAX, 1mL s.c. injection, 3 vaccinations, days 0, 7 and 28
  Arms: JE-VAX

SUMMARY:
The objective is to demonstrate the non-inferiority of the Japanese Encephalitis vaccine IC51 compared to JE-VAX in healthy subjects aged > or = 18 years

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Written informed consent obtained prior to study entry

Exclusion Criteria:

* History of clinical manifestation of any flavivirus infection
* History of vaccination against Japanese encephalitis (JE), Yellow fever and Dengue fever (an anti-JEV neutralizing antibody titer >= 1:10 at baseline is acceptable for inclusion, these subjects will be part of the safety population, but will not be analyzed for immunogenicity in the per-protocol analysis)
* Use of any other investigational or non-registered drug or vaccine in addition to the study vaccine during the study period or within 30 days preceding the first dose of study vaccine
* Immunodeficiency including post-organ-transplantation or immunosuppressive therapy
* A family history of congenital or hereditary immunodeficiency
* History of autoimmune disease
* Any acute infections within 4 weeks prior to enrollment
* Infection with HIV, Hepatitis B or Hepatitis C
* Pregnancy, lactation or unreliable contraception in female subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 867 (Actual)
Dates: Start 2005-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Kaltenboeck, Ph.D., Study Director — Valneva Austria GmbH

RESULTS

PARTICIPANT FLOW:
Groups:
- IC51: IC51
- JE-VAX: JE-VAX
Period: Overall Study
Arm/Group | IC51 | JE-VAX
Started | 430 | 437
Completed | 399 | 397
Not Completed | 31 | 40
Not completed — Withdrawal by Subject | 9 | 10
Not completed — Protocol Violation | 2 | 8
Not completed — Lost to Follow-up | 5 | 5
Not completed — administrative reasons | 9 | 11
Not completed — Adverse Event | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IC51 | JE-VAX | Total
Number analyzed (Participants) | 430 | 437 | 867
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (14.5) | 41.1 (14.4) | 41.3 (14.4)
Sex/Gender, Customized [Number; unit: participants]
  Female | 267 | 258 | 525
  Male | 161 | 177 | 338
  Unknown | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Europe | 100 | 103 | 203
  North America | 330 | 334 | 664

OUTCOME MEASURES:

1. Primary Outcome: SCR (Seroconversion Rate)of IC51 Compared to JE-VAX at Day 56
Description: SCR: anti-JEV neutralizing antibody titer ≥1:10
Time Frame: Day 56
Population: Per Protocol Population: all randomized subjects without any protocol deviations as defined in the Statistical Analysis Plan
Measure: Number; unit: percentage of participants
Arm/Group | IC51 | JE-VAX
Number analyzed (Participants) | 365 | 370
percentage of participants | 96.4 | 93.6

2. Secondary Outcome: Safety and Adverse Events
Time Frame: until Day 56
Reporting Status: Not Posted

3. Secondary Outcome: Immunogenicity at Day 28
Time Frame: Day 28
Reporting Status: Not Posted

4. Secondary Outcome: Immunogenicity at Day 56 for North America vs. Europe
Time Frame: Day 56
Reporting Status: Not Posted

5. Secondary Outcome: Immunogenicity at Day 56 for Subjects Older vs. Younger Than 50 Years of Age
Time Frame: Day 56
Reporting Status: Not Posted

6. Primary Outcome: GMT (Geometric Mean Titer) of IC51 Compared to JE-VAX at Day 56
Description: GMT: geometric mean of PRNT50
Time Frame: Day 56
Population: PP Population: All randomized subjects without any major protocol deviations as assessed during a Data Review Meeting. Subjects who were randomized incorrectly or took the wrong study medications were also excluded.
Measure: Geometric Mean (Standard Deviation); unit: titers
Arm/Group | IC51 | JE-VAX
Number analyzed (Participants) | 361 | 364
titers | 243.6 (1163.1) | 102 (221)

ADVERSE EVENTS:
Description: numbers provided for safety population (N= 863)
Arm/Group | IC51 | JE-VAX
Serious Adverse Events (participants affected / at risk) | 1/428 | 0/435
Other Adverse Events (participants affected / at risk) | 217/428 | 213/435
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IC51 (N=428) | JE-VAX (N=435)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IC51 (N=428) | JE-VAX (N=435)
Nausea (Gastrointestinal disorders) | 29 | 39
Fatigue (General disorders) | 54 | 48
Influenza like Ilness (General disorders) | 54 | 55
Pyrexia (General disorders) | 24 | 21
Nasopharyngitis (Infections and infestations) | 26 | 33
Myalgia (Musculoskeletal and connective tissue disorders) | 88 | 69
Headache (Nervous system disorders) | 113 | 125
Diarrhoea (Gastrointestinal disorders) | 7 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 11
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 12 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other